CLINICAL TRIAL: NCT02773849
Title: A Phase III, Open Label Study to Evaluate the Safety and Efficacy of INSTILADRIN® (rAd-IFN)/Syn3) Administered Intravesically to Patients With High-Grade, BCG Unresponsive Non-Muscle Invasive Bladder Cancer (NMIBC)
Brief Title: ADSTILADRIN (=INSTILADRIN) in Patients With High-Grade, Bacillus Calmette-Guerin (BCG) Unresponsive Non-Muscle Invasive Bladder Cancer (NMIBC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Collaborators: FKD Therapies Oy (Industry); Society of Urologic Oncology Clinical Trials Consortium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rAd-IFN-CS-003; 000418 (Other: Ferring)
Record Dates: First submitted 2016-04-19; First posted 2016-05-16 (Estimated); Results first posted 2022-07-13 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Superficial Bladder Cancer
Keywords: IFN; BCG-unresponsive; Non-Muscle Invasive Bladder Cancer (NMIBC)
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- ADSTILADRIN (Experimental): Intravesical administration of ADSTILADRIN into the bladder
  Interventions: Biological: ADSTILADRIN

INTERVENTIONS:
Biological: ADSTILADRIN
  Other Names: rAd-IFN/SYN3NODA; INSTILADRIN

SUMMARY:
Previous multi-dose Phase I and Phase II clinical studies have demonstrated that ADSTILADRIN is a safe and effective treatment for BCG-refractory and recurrent NMIBC. This Phase III study is designed to expand those observations using a high dose of ADSTILADRIN in patients that are "BCG Unresponsive" which refers to patients with high-grade NMIBC who are unlikely to benefit from and should not receive further intravesical BCG.

DETAILED DESCRIPTION:
Recombinant IFN alpha2b has pleiotropic effects that contribute to antitumor activity in Non-Muscle Invasive Bladder Cancer (NMIBC). ADSTILADRIN is a non-replicating adenovirus vector harboring the human IFN alpha2b gene. When combined with the excipient Syn3, intravesical administration of the rAd-IFN results in transduction of the virus into the epithelial cell lining in the bladder. The IFN alpha2b gene is incorporated into the cellular DNA resulting in the synthesis and expression of large amounts of IFN alpha2b protein. Clinical studies have confirmed that IFN alpha2b protein can be measured in the urine of patients treated with ADSTILADRIN within 24 hours after dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older at the time of consent
2. Able to give informed consent
3. Had, at entry, confirmed by a pathology report:

   Carcinoma in situ (CIS) only; Ta/T1 high-grade disease with concomitant CIS; or Ta/T1 high-grade disease without concomitant CIS
4. Are "BCG Unresponsive" which refers to patients with high-grade NMIBC who were unlikely to benefit from and who did not receive further intravesical BCG. The term "BCG unresponsive" included patients who did not respond to BCG treatment and had a persistent high-grade recurrence within 12 months after BCG was initiated, and those who despite an initial complete response (CR) to BCG, relapsed with high-grade CIS within 12 months of their last intravesical treatment with BCG or relapsed with high-grade Ta/T1 NMIBC within 6 months of their last intravesical treatment with BCG. The following criteria defined the patients who were eligible for inclusion in the study:

   * Had received at least 2 previous courses of BCG within a 12 month period. This was defined as at least 5 of 6 induction BCG instillations and at least 2 out of 3 instillations of maintenance BCG, or at least 2 of 6 instillations of a second induction course, where maintenance BCG was not given;

     * Exception: those who had T1 high-grade disease at first evaluation after induction BCG alone (at least 5 of 6 doses) qualified in the absence of disease progression.
   * At the time of tumor recurrence, patients with CIS alone or high-grade Ta/T1 with CIS were within 12 months of last exposure to BCG and patients with high-grade Ta/T1 without CIS were within 6 months of last exposure to BCG;
   * No maximum limit to the amount of BCG administered; and
   * All visible papillary tumors were required to be resected and those with persistent T1 disease on transurethral resection of bladder tumor (TURBT) underwent an additional re-TURBT within 14 to 60 days prior to beginning study treatment. Obvious areas of CIS should also be fulgurated.
5. Available for the whole duration of the study
6. Life expectancy >2 years, in the opinion of the investigator
7. Eastern Cooperative Oncology Group (ECOG) status 2 or less
8. Absence of concomitant upper tract urothelial carcinoma or urothelial carcinoma within the prostatic urethra. Freedom from upper tract disease (if clinically indicated) as indicated by no evidence of upper tract tumor by either intravenous pyelogram, retrograde pyelogram, computed tomography (CT) scan with or without urogram, or magnetic resonance imaging (MRI) with or without urogram performed within 6 months of enrollment
9. Patients with prostate cancer on active surveillance at low risk for progression, defined as Prostate-Specific Antigen (PSA) < 10 ng/dL, Gleason score 6 and clinical stage tumor-1 (cT1) were permitted to be in the study at the discretion of the investigator (see exclusion criterion 10).
10. Female patients of childbearing potential were required to use maximally effective birth control during the period of therapy, were required to use contraception for 1 month following the last study drug infusion and were required to have a negative urine or serum pregnancy test upon entry into this study. Otherwise, female patients were required to be postmenopausal (no menstrual period for a minimum of 12 months) or surgically sterile. 'Maximally effective birth control' meant that the patient, if sexually active, used a combination of two methods of birth control that were approved and recognized to be effective by Regulatory Agencies
11. Male patients were required to be surgically sterile or willing to use a double barrier contraception method upon enrollment, during the course of the study, and for 1 month following the last study drug infusion; and
12. Adequate lab values

Exclusion Criteria:

1. Current or previous evidence of muscle invasive (muscularis propria) or metastatic disease presented at the screening visit. Examples of increased risk of metastatic disease included (but were not limited to):

   * Presence of lymphovascular invasion and/micropapillary disease as shown in the histology of the biopsy sample; and
   * Patients with T1 disease accompanied by the presence of hydronephrosis secondary to the primary tumor
2. Current systemic therapy for bladder cancer
3. Current or prior pelvic external beam radiotherapy within 5 years of entry
4. Prior treatment with adenovirus-based drugs
5. Suspected hypersensitivity to IFN alfa2b
6. Symptomatic urinary tract infection or bacterial cystitis (once satisfactorily treated, patients could have entered the study)
7. Clinically significant and unexplained elevated liver or renal function tests
8. Women who were pregnant or lactating or refused to commit to use contraception throughout the study
9. Any other significant disease or other clinical findings which, in the opinion of the investigator, prevented study entry
10. History of malignancy of another organ system within the past 5 years, except treated basal cell carcinoma or squamous cell carcinoma of the skin and ≤ pathological tumor-2 (pT2) upper tract urothelial carcinoma at least 24 months after nephroureterectomy. Also patients with genitourinary cancers other than urothelial cancer or prostate cancer that were under active surveillance were excluded (see inclusion criterion 9)
11. Patients who could not hold instillation for 1 hour
12. Patients who could not tolerate intravesical dosing or intravesical surgical manipulation; and
13. Intravesical therapy within 8 weeks prior to beginning study treatment with the exception of:

    * cytotoxic agents (e.g. Mitomycin C, doxorubicin and epirubicin) when administered as a single instillation immediately following a TURBT procedure which was permitted between 14 to 60 days prior to beginning study treatment
    * previous intravesical BCG therapy, which could be given at least 5 weeks before the diagnostic biopsy required for entry into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2023-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Boorjian, MD, Principal Investigator — Mayo Clinic
Locations (34):
- United States (34):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Keck School of Medicine at USC Medical Center, Los Angeles, California
  - The Urology Center of Colorado, Denver, Colorado
  - University of Florida - UF Health Davis Center Pavilion and Shands Med Plaza, Gainesville, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Chicago - Comprehensive Cancer Research Center, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Johns Hopkins Kimmel Cancer Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Spectrum Health Medical Group, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Delaware Valley Urology, LLC, Voorhees Township, New Jersey
  - SUNY Upstate Medical Center, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina (UNC) - Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Regional Urology, Greenville, South Carolina
  - Carolina Urologic research Center, Myrtle Beach, South Carolina
  - Vanderbilt University Medical Center Dept. of Urologic Surgery, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - The Univ. of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Urology of Virginia, Virginia Beach, Virginia
  - West Virginia University Cancer Institute, Morgantown, West Virginia
  - University of Wisconsin - Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Boorjian SA, Alemozaffar M, Konety BR, Shore ND, Gomella LG, Kamat AM, Bivalacqua TJ, Montgomery JS, Lerner SP, Busby JE, Poch M, Crispen PL, Steinberg GD, Schuckman AK, Downs TM, Svatek RS, Mashni J Jr, Lane BR, Guzzo TJ, Bratslavsky G, Karsh LI, Woods ME, Brown G, Canter D, Luchey A, Lotan Y, Krupski T, Inman BA, Williams MB, Cookson MS, Keegan KA, Andriole GL Jr, Sankin AI, Boyd A, O'Donnell MA, Sawutz D, Philipson R, Coll R, Narayan VM, Treasure FP, Yla-Herttuala S, Parker NR, Dinney CPN. Intravesical nadofaragene firadenovec gene therapy for BCG-unresponsive non-muscle-invasive bladder cancer: a single-arm, open-label, repeat-dose clinical trial. Lancet Oncol. 2021 Jan;22(1):107-117. doi: 10.1016/S1470-2045(20)30540-4. Epub 2020 Nov 27. PMID 33253641
- [Derived] Konety BR, Lotan Y, Myers A. Safety of nadofaragene firadenovec-vncg: review of data from phase 2 and phase 3 studies. Can J Urol. 2025 Mar 18;32(1):29-36. doi: 10.32604/cju.2025.064710. PMID 40194933

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled in the study who had at entry, confirmed by a pathology report: CIS only or Ta/T1 high- grade disease with concomitant CIS, or Ta/T1 high-grade disease without concomitant CIS and were "BCG unresponsive" which referred to patients with high-grade NMIBC who were unlikely to benefit from and who did not receive further intravesical BCG.
Period: Overall Study
Arm/Group | ADSTILADRIN
Started | 157
Completed | 95
Not Completed | 62
Not completed — Lost to Follow-up | 11
Not completed — Death | 26
Not completed — Withdrawal by Subject | 5
Not completed — Withdrawal of Consent | 9
Not completed — Other: not due to lack of tolerability | 11

BASELINE CHARACTERISTICS:
Groups:
- Carcinoma in Situ: Patients with Carcinoma in situ (CIS) with or without concomitant high-grade Ta or T1 papillary disease
- Papillary Disease: Patients with high-grade Ta or T1 papillary disease (without concomitant CIS)
- Total: Total of all reporting groups
Arm/Group | Carcinoma in Situ | Papillary Disease | Total
Number analyzed (Participants) | 107 | 50 | 157
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 13 | 38
  >=65 years | 82 | 37 | 119
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 28
  Male | 95 | 34 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 99 | 49 | 148
  Unknown or Not Reported | 5 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 99 | 47 | 146
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 107 | 50 | 157
Height [Mean (Standard Deviation); unit: cm] | 174.7 (9.8) | 170.9 (10.3) | 173.5 (10.1)
Weight [Mean (Standard Deviation); unit: kg] | 90.14 (20.9) | 85.88 (18.6) | 88.78 (20.2)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.38 (5.7) | 29.28 (5.1) | 29.34 (5.5)
ECOG Status [Count of Participants; unit: Participants] — The ECOG performance status was assessed according to a scale from 0 to 5, where 0 is fully active, able to carry on all pre-disease performance without restriction and where 4 is completely disabled, cannot carry on any self-care, totally confined to bed or chair and 5 is dead.
  Participants
    Total ECOG of 0 | 97 | 43 | 140
    Total ECOG of 1 | 7 | 6 | 13
    Total ECOG of 2 | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Complete Response Rate Based on Patients With Carcinoma in Situ (CIS), With or Without Concomitant High-grade Ta or T1 Papillary Disease.
Description: A patient in the CIS cohort was judged to have achieved CR where urine cytology was reported as normal, atypical, degenerative, reactive, inflammatory, or nonspecific AND cystoscopy was reported as normal or with findings that did not include evidence of low-grade or high-grade recurrence. Bladder biopsy, if performed (not mandatory), demonstrated an absence of low-grade or high-grade recurrence.
Time Frame: 12 Months
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- Carcinoma in Situ: CIS participants had at entry, confirmed by a pathology report: Carcinoma in situ (CIS) only or Ta/T1 highgrade disease with concomitant CIS AND were "BCG unresponsive" which referred to patients with highgrade NMIBC who were unlikely to benefit from and who did not receive further intravesical BCG. The term "BCG unresponsive" included patients who did not respond to BCG treatment and had a persistent high-grade recurrence within 12 months after BCG was initiated, and those who, despite an initial CR to BCG, relapsed with CIS within 12 months of their last intravesical treatment with BCG or relapsed with high-grade Ta/T1 NMIBC within 6 months of their last intravesical treatment with BCG.
Arm/Group | Carcinoma in Situ
Number analyzed (Participants) | 103
participants | 55 [43.3 to 63.3]

2. Secondary Outcome: Durability of Complete Response in Patients With CIS (With or Without Concomitant Ta or T1 Papillary Disease) Who Achieve a Complete Response.
Description: Durability of complete response (CR) was defined as the time from first observed CR to the documented treatment failure. Patients without treatment failure were censored at the last disease assessment not showing treatment failure, where treatment failure was defined as high-grade disease recurrence, disease progression, or death, whichever occurred earlier.
Time Frame: Up to 57 months
Population: Patients who achieved CR
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carcinoma in Situ
Number analyzed (Participants) | 55
Months | 9.72 [9.17 to 23.95]

3. Secondary Outcome: Rate of Event-free Survival, Where Event-free Survival is Defined as High-grade Recurrence Free (HGRF) Survival in Patients With High-grade Ta or T1 Disease (Without Concomitant CIS)
Description: Complete response rate will be measured by determining the number of patients without recurrence of high-grade disease using results from urine cytology, cystoscopy, and biopsy of the bladder. Incidence of HGRF survival at Months 3, 6, 9, and 12, and every 3 months up to Month 24, and then at Months 36, 48, and 57.
Time Frame: up to 57 months
Population: A patient was judged to have achieved HGRF survival at a time point (eg, Months 3, 6, 9, and 12) if the patient was alive and without documented recurrence of high-grade disease or muscle-invasive disease progression as assessed by the Investigator at that time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Papillary Disease
Number analyzed (Participants) | 48
Participants
  Month 3 | 35
  Month 6 | 30
  Month 9 | 28
  Month 12 | 21
  Month 24 | 16
  Month 36 | 11
  Month 48 | 7
  Month 57 | 7

4. Secondary Outcome: Durability of High-grade-recurrence-free Survival in Patients With High-grade Ta or T1 Papillary Disease (With or Without Concomitant CIS)
Description: HGRF survival was defined as the time from the first dose to the first recurrence of high-grade disease (including muscle-invasive disease progression and death due to any cause). Patients without high-grade disease recurrence were censored at the last disease assessment not showing high-grade disease recurrence.
Time Frame: Up to 57 months
Population: Patients with no recurrence of high-grade disease
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Total: All Patients
Arm/Group | Carcinoma in Situ | Papillary Disease | Total
Number analyzed (Participants) | 103 | 48 | 151
Months
  HGRF Survival | 5.95 [3.38 to 8.31] | 12.35 [6.67 to 20.27] | 7.31 [5.68 to 11.93]
  Probability of duration of HGRF survival for 57 months | 13.2 [6.9 to 21.5] | 32.7 [19.5 to 46.6] | 19.0 [12.6 to 26.4]
  Probability of duration of HGRF survival for 48 months | 16.7 [10.1 to 24.9] | 32.7 [19.5 to 46.6] | 21.6 [15.2 to 28.8]
  Probability of duration of HGRF survival for 36 months | 19.3 [12.2 to 27.6] | 32.7 [19.5 to 46.6] | 23.6 [17.0 to 30.8]

5. Secondary Outcome: Incidence of Cystectomy at 12 Months, 2 Years and 5 Years
Description: The incidence of cystectomy is described as the proportion of patients undergoing radical cystectomy for any reason after the first dose, within 12 months, 2 years and 5 years.
Time Frame: 60 Months
Population: Proportion of patients undergoing cystectomy within 5 years, 2 years and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Carcinoma in Situ | Papillary Disease | Total
Number analyzed (Participants) | 103 | 48 | 151
Participants
  12 months | 27 | 7 | 34
  2 years | 35 | 10 | 45
  5 years | 42 | 14 | 56

6. Secondary Outcome: Overall Survival Rate in All Patients
Description: Overall survival rate was defined as the time from the first dose to death due to any cause. Patients who were still alive were censored at the last date the patient was known to be alive. Overall survival rate is a Kaplan-Meier estimate of the survivor function at each specific time point. The 95% CI is calculated using the Greenwood's formula with a log-log transformation. Percentage is calculated using the number of patients in the column heading as the denominator.
Time Frame: 60 Months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Carcinoma in Situ | Papillary Disease | Total
Number analyzed (Participants) | 103 | 48 | 151
percentage of patients
  3 months | 100 [NA to NA] — 95% confidence interval could not be calculated due to an insufficient number of participants with events | 100 [NA to NA] — 95% confidence interval could not be calculated due to an insufficient number of participants with events | 100 [NA to NA] — 95% confidence interval could not be calculated due to an insufficient number of participants with events
  6 months | 99 [93.0 to 99.9] | 100 [NA to NA] — 95% confidence interval could not be calculated due to an insufficient number of participants with events | 99.3 [95.3 to 99.9]
  9 months | 98 [92.2 to 99.5] | 100 [NA to NA] — 95% confidence interval could not be calculated due to an insufficient number of participants with events | 98.6 [94.7 to 99.7]
  12 months | 98 [92.2 to 99.5] | 97.9 [85.8 to 99.7] | 98 [93.8 to 99.3]
  24 months | 94.9 [88.1 to 97.8] | 93.5 [81.2 to 97.9] | 94.5 [89.2 to 97.2]
  48 months | 83.6 [74.3 to 89.8] | 88.9 [75.4 to 95.3] | 85.4 [78.3 to 90.3]
  60 months | 76.3 [64.6 to 84.5] | 85.9 [70.9 to 93.5] | 79.7 [71.0 to 86.0]

7. Secondary Outcome: Anti-adenoviral Antibody Levels for Correlation to Response Rate
Description: Measurement of anti-adenoviral antibody levels at each dosing period, withdrawal, and at 12 months were done. A patient was considered to have a positive immunogenic response in anti-adenoviral antibodies if a post-baseline titration demonstrated a greater than a 2-fold dilution increase from baseline.
  The table represent data at any time during the 12 months period, which means that the patients were included in the Yes group if they at any measurement during the trial had a 2-fold dilution increase from baseline.
Time Frame: 12 Months
Population: Patients with Positive Immunogenic Response in Anti-Adenoviral Antibodies at Post-Baseline based on patients who had achieved High-Grade Recurrence Free Survival at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Carcinoma in Situ | Papillary Disease | Total
Number analyzed (Participants) | 89 | 45 | 134
Participants
  Yes | 63 | 34 | 97
  No | 26 | 11 | 37

8. Secondary Outcome: Safety of ADSTILADRIN
Description: The type, incidence, relatedness and severity of treatment emergent adverse events of ADSTILADRIN as assessed by NCI-CTCAE V4.03 were monitored.
Time Frame: 60 Months
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Carcinoma in Situ | Papillary Disease | Total
Number analyzed (Participants) | 107 | 50 | 157
Participants
  TEAE | 101 | 45 | 146
  Serious TEAE | 10 | 9 | 19
  NCI-CTCAE Grade 3/4/5 TEAE | 22 | 12 | 34

9. Secondary Outcome: Durability of Response During the Long-term Follow-up Period.
Description: Durability will be measured by determining the number of patients without recurrence of high-grade disease using results from urine cytology, cystoscopy, and biopsy of the bladder if clinically indicated.
Time Frame: Up to 60 Months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carcinoma in Situ | Papillary Disease | Total
Number analyzed (Participants) | 107 | 50 | 157
months | 48.92 [37.88 to 59.47] | 59.01 [46.55 to 60.52] | 50.83 [39.10 to 60.02]

ADVERSE EVENTS:
Time Frame: 60 months
Description: The Month 60 final dataset was used for all Adverse Event Reporting data.
Groups:
- Carcinoma in Situ (CIS): Patients had at entry, confirmed by a pathology report: Carcinoma in situ (CIS) only or Ta/T1 high-grade disease with concomitant CIS and were "BCG unresponsive" which referred to patients with high-grade NMIBC who were unlikely to benefit from and who did not receive further intravesical BCG. The term "BCG unresponsive" included patients who did not respond to BCG treatment and had a persistent high-grade recurrence within 12 months after BCG was initiated, and those who, despite an initial CR to BCG, relapsed with CIS within 12 months of their last intravesical treatment with BCG or relapsed with high-grade Ta/T1 NMIBC within 6 months of their last intravesical treatment with BCG.
- Papillary Disease (Without Concomitant CIS): Patients had at entry, confirmed by a pathology report Ta/T1 high-grade disease without concomitant CIS and were "BCG unresponsive" which referred to patients with high-grade NMIBC who were unlikely to benefit from and who did not receive further intravesical BCG. The term "BCG unresponsive" included patients who did not respond to BCG treatment and had a persistent high-grade recurrence within 12 months after BCG was initiated, and those who, despite an initial CR to BCG, relapsed with high-grade Ta/T1 high-grade disease without concomitant CIS within 12 months of their last intravesical treatment with BCG or relapsed with high- grade Ta/T1 NMIBC within 6 months of their last intravesical treatment with BCG.
- Total TEAE: Total Treatment-Emergent Adverse Events (TEAE) in the Study.
Arm/Group | Carcinoma in Situ (CIS) | Papillary Disease (Without Concomitant CIS) | Total TEAE
All-Cause Mortality (participants affected / at risk) | 21/107 | 5/50 | 26/157
Serious Adverse Events (participants affected / at risk) | 10/107 | 9/50 | 19/157
Other Adverse Events (participants affected / at risk) | 101/107 | 45/50 | 146/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carcinoma in Situ (CIS) (N=107) | Papillary Disease (Without Concomitant CIS) (N=50) | Total TEAE (N=157)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (2) | 1 (2)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Translational cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carcinoma in Situ (CIS) (N=107) | Papillary Disease (Without Concomitant CIS) (N=50) | Total TEAE (N=157)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 5 (5) | 7 (7)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 7 (7) | 17 (17)
Nausea (Gastrointestinal disorders) | 8 (8) | 4 (4) | 12 (12)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3) | 6 (6)
Chills (General disorders) | 18 (18) | 6 (6) | 24 (24)
Fatigue (General disorders) | 29 (29) | 8 (8) | 37 (37)
Influenza like illness (General disorders) | 4 (4) | 4 (4) | 8 (8)
Instillation site discharge (General disorders) | 37 (37) | 15 (15) | 52 (52)
Malaise (General disorders) | 2 (2) | 4 (4) | 6 (6)
Pain (General disorders) | 9 (9) | 2 (2) | 11 (11)
Pyrexia (General disorders) | 18 (18) | 7 (7) | 25 (25)
Bronchitis (Infections and infestations) | 1 (1) | 5 (5) | 6 (6)
Nasopharyngitis (Infections and infestations) | 8 (8) | 2 (2) | 10 (10)
Sinusitus (Infections and infestations) | 3 (3) | 3 (3) | 6 (6)
Urinary tract infection (Infections and infestations) | 11 (11) | 12 (12) | 23 (23)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4) | 10 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 8 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (5) | 12 (12)
Dizziness (Nervous system disorders) | 8 (8) | 6 (6) | 14 (14)
Headache (Nervous system disorders) | 16 (16) | 8 (8) | 24 (24)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 3 (3) | 4 (4)
Bladder pain (Renal and urinary disorders) | 9 (9) | 3 (3) | 12 (12)
Bladder spasm (Renal and urinary disorders) | 22 (22) | 9 (9) | 31 (31)
Dysuria (Renal and urinary disorders) | 17 (17) | 8 (8) | 25 (25)
Haematuria (Renal and urinary disorders) | 19 (19) | 7 (7) | 26 (26)
Micturition urgency (Renal and urinary disorders) | 20 (20) | 9 (9) | 29 (29)
Pollakiuria (Renal and urinary disorders) | 9 (9) | 6 (6) | 15 (15)
Urinary incontinence (Renal and urinary disorders) | 8 (8) | 1 (1) | 9 (9)
Hypertension (Vascular disorders) | 8 (8) | 3 (3) | 11 (11)
Nocturia (Renal and urinary disorders) | 4 (4) | 3 (3) | 7 (7)
Urinary retention (Renal and urinary disorders) | 4 (4) | 3 (3) | 7 (7)
Procedural pain (Injury, poisoning and procedural complications) | 6 (6) | 1 (1) | 7 (7)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT02773849/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/49/NCT02773849/SAP_001.pdf